CLINICAL TRIAL: NCT06656637
Title: To Drill or Not to Drill: Do Memory Drills Help Strengthen Prospective Memory and Decrease Veterans' Concerns About Prospective Memory Problems?
Brief Title: To Drill or Not to Drill: Do Memory Drills Help Train the Ability to "Remember to Remember" in Veterans
Acronym: PMIS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Delany Thrasher, Director of Neuropsychology, Health Sciences Assistant Clinical Professer, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-24-0693
Record Dates: First submitted 2024-10-17; First posted 2024-10-24 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Memory Deficit
Keywords: Prospective memory; Memory intervention; Memory drilling; Veterans; Memory concerns; Compensatory strategies; Cognitive training
MeSH Terms: conditions — Memory Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Memory Drilling BRAIN ITP (EXP) (Experimental): In the BRAIN ITP, the standard PM training for both the experimental (EXP) and control group (CON1), takes place during the patient's individual cognitive training sessions with the cognitive trainer. In total, there are seven sessions. At each of these sessions the cognitive trainer will review a new compensatory strategy for PM and assign a naturalistic PM practice task as homework to practice the strategy. The experimental group will receive the additional computerized "memory drills" training.
- Standard of Care BRAIN ITP (CON1) (Active Comparator): In the BRAIN ITP, the standard PM training for both the experimental (EXP) and control group (CON1), takes place during the patient's individual cognitive training sessions with the cognitive trainer. In total, there are seven sessions. At each of these sessions the cognitive trainer will review a new compensatory strategy for PM and assign a naturalistic PM practice task as homework to practice the strategy. The CON1 group will not receive the additional memory drilling.
  Interventions: Behavioral: Compensatory Strategies
- Standard of Care PTSD ITP (CON2) (Active Comparator): The PTSD ITP group (CON2) will receive the traditional standard of care (cognitive training and cognitive processing therapy). There is no spaced training or practice.
  Interventions: Behavioral: Compensatory Strategies; Behavioral: Cognitive Processing Therapy

INTERVENTIONS:
Behavioral: Memory Drilling — The experimental group will receive the additional intervention during their seven sessions with their care providers. The intervention is computerized "memory drills" training. This training includes the completion of a list learning memory task (HVLT) and then a PM practice task conducted on the computer at each session.
Behavioral: Compensatory Strategies — Participants learn compensatory strategies to assist with their memory performance. This involves both external strategies, such as calendering and setting alarms, and internal strategies, like imagery and mnemonics.
  Arms: Standard of Care BRAIN ITP (CON1); Standard of Care PTSD ITP (CON2)
Behavioral: Cognitive Processing Therapy — This is PTSD-targeted therapy.
  Arms: Standard of Care PTSD ITP (CON2)

SUMMARY:
The goal of this clinical trial is to memory drilling works in improving the ability to remember to do something later in treatment-seeking veterans. The main question it aims to answer is:

Does adding memory drilling to intensive treatment programs improve the patient's ability to remember to do something later?

Researchers will compare typical standardized memory training to the memory training with drilling to see if drilling improves the veterans' ability to remember tasks they are supposed to do later.

Participants will:

* complete the Operation Mend intensive treatment program with either standard care (either with or without Post-Traumatic Stress Disorder [PTSD] focused trauma therapy) or standard care + memory drilling
* complete a virtual memory assessment at entrance, exit, and three months post exit. This assessment will include questionnaires, interviews, and computerized and naturalistic memory tasks.

DETAILED DESCRIPTION:
Treatment-seeking veterans who come for diagnostics and/or treatment to University of California, Los Angeles (UCLA) Operation Mend show a high level of memory concern. To address this issue, the veterans receive training in evidence-informed compensatory strategies. However, a high level of memory concern remains, and this study aims to investigate the efficacy of adding memory drills to the treatment program.

There is mixed evidence in the literature about whether memory drills, which tend to show improvement in computerized cognitive tasks, generalize to naturalistic forms of memory. Specifically, the efficacy of computerized training for prospective memory (PM), perhaps the most naturalistic form of memory, is understudied. The proposed study seeks to answer the question whether adding a computerized "drilling" of retrospective and prospective memory to Operation Mend's Cognitive Training enhances patients' PM performance & reduces their memory concerns.

Study participants will be only be recruited from participants of the Operation Mend Intensive Treatment Programs (ITPs). The BRAIN ITP is a two-week intensive brain health program for patients who may have a history of mild traumatic brain injury and other comorbidities who wish to focus on improving their day-to-day cognitive functioning, maximizing their brain health as well as reducing the impact of other symptoms such as physical pain. It involves cognitive training sessions and meetings with neuropsychologists, neurologists, occupational therapists, dieticians, etc. The PTSD ITP is a two-week intensive therapy and skills training program for patients who wish to focus on evidence-based treatment for PTSD and other psychological and cognitive comorbidities that involves mental health sessions and meetings with psychiatrists, psychologists, neuropsychologists, etc.

This will be a randomized controlled trial with three groups. The experimental group with BRAIN ITP participants will receive the normal standard of care and memory drilling while the BRAIN ITP control group receives only the normal standard of care. The third control group will come from the PTSD ITP who receive normal standard of care plus PTSD treatment. This control group is included because of indications of a connection between PTSD symptomology and PM deficits.

In the BRAIN ITP, the standard PM training for both the experimental and control group takes place during the patient's individual sessions with a neuropsychologist. In total, there are seven sessions. At each of these sessions the neuropsychologist will review a new compensatory strategy for prospective memory and assign a naturalistic task for completion as homework to practice the strategy. The experimental group will receive the additional "memory drills" training. This training includes the completion of a list learning memory task and then a prospective memory task conducted on the computer at each session. The PTSD ITP group will receive the standard of care (cognitive processing therapy and cognitive training).

Participants will be assessed at baseline (before entering the program), at exit (immediately after the two-week program) and at 3 months post exit. The assessments consist of surveys regarding their PM performance in their day-to-day lives, a computerized and naturalistic objective measurement of PM. All assessments, except for the exit assessment which does not include the naturalistic task, will be administered via Zoom by study staff. Participants will fill out the exit assessment by themselves. The total study time will be approximately 2 to 3.5 hours over the course of approximately 15 to 17 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Only patients that are already accepted and scheduled to participate in an Operation Mend BRAIN Intensive Treatment Program and PTSD Intensive Treatment Program are eligible to participate in the study.

Exclusion Criteria:

* Patients with acute substance abuse disorders are not accepted into Operation Mend programs and are therefore excluded from the study.
* For logistical reasons, patients who are scheduled for arrival at the ITP sooner than 2.5 or 3 weeks are not eligible to participate.
* Patients who do not have tablet, iPad, or computer access are not eligible to participate due to the technical requirements of the computer-based assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Prospective Memory Concerns Questionnaire (PMCQ) | Day 10 of program, three month follow up
  The Prospective Memory Concerns Questionnaire (PMCQ) is a self-report that includes 3 subscales (Forgetting Behaviors, Memory Concerns, Retrieval Failures) and an event-based prospective memory task where they have to remember to write their handedness in the textbox at the end of the questionnaire. It is meant to assess participants experience with prospective memory tasks in their day to day lives. Item scores range from 0 to 3. Total score Range 0 to 105. Higher scores indicate more prospective memory concerns.
Adapted Royal Prince Alfred Prospective Memory Test | three month follow up
  This is a slightly adapted version (ie. using emails instead of posting letters, etc.) of the Royal Prince Alfred Prospective Memory Assessment. It is a lab based but still naturalistic assessment of prospective memory. It involves short term and long term, time and event based prospective memory tasks.
  Total score range 0 to 12. Higher scores indicate better prospective memory performance.
Computerized Prospective Memory Assessment (C-PMAT) | Day 10 of program, three month follow-up
  This is a two-part computerized task that will take no more than 25 minutes total. There are two components to the task: the "ongoing" task and the embedded prospective memory task. The ongoing task will be the same for both parts of the task - a letter 2 back. The first part of the task will involve an event-based prospective memory response while the second part will require a time-based prospective memory response. For the event-based part, participants are told to press the letter "N" itself, instead of the "2 back" button of the ongoing task, when the letter "N" is on the screen. In the time-based part, participants will be told to check the time every 100 seconds while completing the ongoing task. There will be 5 total embedded prospective tasks in each part.
  Total score range is 0 to 10. Higher scores indicate better performance.

SECONDARY OUTCOMES:
Metacognitive Prospective Memory Inventory (MPMI-s) | three month follow-up
  This self-report questionnaire assesses the use of internal and external strategies to assist with memory. It will be used to assess whether the treatment program increased the use of compensatory strategies for prospective memory tasks.
  Total score ranges from 22 - 110. Higher scores reflect better PM abilities.
Cognitive Confidence subscale of MCQ-30 | three month follow-up
  This is a 6-item self report subscale that assesses the patient's confidence/trust in their memory abilities. It will be used to assess patients belief in their memory abilities before and after the program. Total score ranges from 6 to 24. Higher scores indicate worse confidence.
Post-concussive Catastrophizing Scale - cognitive symptoms (PCS-CS) | Day 10 of program, three month follow-up
  This measure is the post concussive catastrophizing scale with a focus on only cognitive symptoms. This will be used to assess if there is a change in the catastrophizing of cognitive abilities in the veteran pre and post treatment. Total score ranges from 0 to 52. Higher scores indicate higher catastrophizing.

CONTACTS AND LOCATIONS:
Overall Officials: Delany Thrasher, PhD, Principal Investigator — University of California, Los Angeles; Kevin Bickart, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
UCLA Health Operation Mend is a comparably small treatment program; the program does not wish to share any IPD from research participants because their research participation is contingent on receiving treatment at the organization. No individual participant data will be shared.

REFERENCES:
- [Background] Wijenberg MLM, Hicks AJ, Downing MG, van Heugten CM, Stapert SZ, Ponsford JL. Relevance of the Fear-Avoidance Model for Chronic Disability after Traumatic Brain Injury. J Neurotrauma. 2020 Dec 15;37(24):2639-2646. doi: 10.1089/neu.2020.7135. Epub 2020 Sep 22. PMID 32842860
- [Background] Wells A, Cartwright-Hatton S. A short form of the metacognitions questionnaire: properties of the MCQ-30. Behav Res Ther. 2004 Apr;42(4):385-96. doi: 10.1016/S0005-7967(03)00147-5. PMID 14998733
- [Background] Radford KA, Lah S, Say MJ, Miller LA. Validation of a new measure of prospective memory: the Royal Prince Alfred Prospective Memory Test. Clin Neuropsychol. 2011 Jan;25(1):127-40. doi: 10.1080/13854046.2010.529463. Epub 2010 Nov 19. PMID 21108144
- [Background] Sugden N, Thomas M, Kiernan M, Wilesmith M. Validation of the Prospective Memory Concerns Questionnaire (PMCQ). Front Hum Neurosci. 2021 Aug 26;15:686850. doi: 10.3389/fnhum.2021.686850. eCollection 2021. PMID 34512292
- [Background] Mioni G, Stablum F, McClintock SM, Cantagallo A. Time-based prospective memory in severe traumatic brain injury patients: the involvement of executive functions and time perception. J Int Neuropsychol Soc. 2012 Jul;18(4):697-705. doi: 10.1017/S1355617712000306. Epub 2012 Mar 20. PMID 22433779
- [Background] Sheppard DP, Rau HK, Werhane ML, Fonseca LM, Chaytor NS, Peskind ER, Pagulayan KF. Associations between Intra-Individual Neurocognitive Variability and Prospective Memory in Veterans with Mild Traumatic Brain Injury History and Posttraumatic Stress Disorder. Arch Clin Neuropsychol. 2022 Aug 23;37(6):1221-1227. doi: 10.1093/arclin/acac014. PMID 35470369
- [Background] Rosen AC, Sugiura L, Kramer JH, Whitfield-Gabrieli S, Gabrieli JD. Cognitive training changes hippocampal function in mild cognitive impairment: a pilot study. J Alzheimers Dis. 2011;26 Suppl 3(Suppl 3):349-57. doi: 10.3233/JAD-2011-0009. PMID 21971474
- [Background] Raskin SA, Williams J, Aiken EM. A review of prospective memory in individuals with acquired brain injury. Clin Neuropsychol. 2018 Jul;32(5):891-921. doi: 10.1080/13854046.2018.1455898. Epub 2018 Apr 2. PMID 29609519
- [Background] Pagulayan KF, Rau H, Madathil R, Werhane M, Millard SP, Petrie EC, Parmenter B, Peterson S, Sorg S, Hendrickson R, Mayer C, Meabon JS, Huber BR, Raskind M, Cook DG, Peskind ER. Retrospective and Prospective Memory Among OEF/OIF/OND Veterans With a Self-Reported History of Blast-Related mTBI. J Int Neuropsychol Soc. 2018 Apr;24(4):324-334. doi: 10.1017/S1355617717001217. Epub 2017 Dec 29. PMID 29284552
- [Background] Palermo L, Cinelli MC, Piccardi L, De Felice S, Ciurli P, Incoccia C, Zompanti L, Guariglia C. Cognitive functions underlying prospective memory deficits: A study on traumatic brain injury. Appl Neuropsychol Adult. 2020 Mar-Apr;27(2):158-172. doi: 10.1080/23279095.2018.1501374. Epub 2018 Oct 31. PMID 30380921
- [Background] Coyle H, Traynor V, Solowij N. Computerized and virtual reality cognitive training for individuals at high risk of cognitive decline: systematic review of the literature. Am J Geriatr Psychiatry. 2015 Apr;23(4):335-359. doi: 10.1016/j.jagp.2014.04.009. Epub 2014 May 14. PMID 24998488